CLINICAL TRIAL: NCT04585932
Title: Phase 2 Response Evaluation of Finite Systemic Therapy With Advanced Androgen Signaling Inhibition and Radiation Therapy for Oligorecurrent Prostate Cancer (RESTART)
Brief Title: Androgen Deprivation Therapy and Apalutamide With or Without Radiation Therapy for the Treatment of Biochemically Recurrent Prostate Cancer, RESTART Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: At the request of the ad interim Department Chairman due to PI is no longer at institution.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1093; NCI-2020-02553 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1093 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-05-19; First posted 2020-10-14 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Metastatic Prostate Carcinoma; Oligometastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide; luprolide acetate gel depot; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (apalutamide, leuprolide, degarelix) (Active Comparator): Patients receive apalutamide PO QD on days 1-28 and ADT consisting of leuprolide IM every 12 weeks or degarelix SC every 4 weeks. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Apalutamide; Drug: Degarelix; Drug: Leuprolide Acetate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (apalutamide, leuprolide, degarelix, RT) (Experimental): Patients receive apalutamide PO QD on days 1-28 and ADT consisting of leuprolide IM every 12 weeks or degarelix SC every 4 weeks. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo RT between cycles 4-7 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Apalutamide; Drug: Degarelix; Drug: Leuprolide Acetate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Drug: Degarelix — Given SC
  Other Names: FE200486; Firmagon
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group II (apalutamide, leuprolide, degarelix, RT)

SUMMARY:
This phase II trial studies how well androgen deprivation therapy and apalutamide with or without radiation therapy works for the treatment of prostate cancer that has a rise in the blood level of prostate-specific antigen (PSA) and has come back after treatment with surgery or radiation (biochemically recurrent). Androgens can cause the growth of prostate tumor cells. Apalutamide may help fight prostate cancer by blocking the use of androgens by the tumor cells. Androgen deprivation therapy drugs, leuprolide or degarelix, work to lower the amount of androgen in the body, also preventing the tumor cells from growing. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving radiation therapy with apalutamide and androgen deprivation therapy may help to control prostate cancer that has come back in only a few (up to 5) spots in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess PSA progression-free survival in both treatment arms.

SECONDARY OBJECTIVES:

I. To assess time of recovery of serum testosterone in both treatment arms. II. To assess PSA progression-free survival and overall survival following testosterone recovery in both treatment arms.

III. To assess safety of androgen deprivation therapy (ADT) + apalutamide as well as ADT + apalutamide in combination radiation therapy.

IV. To assess the time to first new metastasis or local / pelvic recurrence in both treatment arms.

V. To assess the impact of both treatment arms on quality of life. VI. To assess the impact of both treatment arms on metabolic syndrome parameters.

VII. To assess the impact of both treatment arms on bone density. VIII. To investigate the association of changes in repeat advanced imaging with outcome.

IX. To compare fluciclovine and prostate specific membrane antigen (PSMA) positron emission tomography (PET)/computed tomography (CT).

EXPLORATORY OBJECTIVE:

I. To identify potential markers of response or resistance to the administered therapies.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive apalutamide orally (PO) once daily (QD) on days 1-28 and ADT consisting of leuprolide intramuscularly (IM) every 12 weeks or degarelix subcutaneously (SC) every 4 weeks. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive apalutamide PO QD on days 1-28 and ADT consisting of leuprolide IM every 12 weeks or degarelix SC every 4 weeks. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy (RT) between cycles 4-7 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* Signed informed consent form (ICF) indicating that the subject understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Consent to MD Anderson laboratory protocol Lab02-152
* Available tumor tissue sample (recently collected +/- archival)
* Biochemically recurrent prostate cancer following definitive treatment with radical prostatectomy or / and external beam radiation therapy. Patient may have received prior androgen deprivation with or without other treatments in the neoadjuvant, adjuvant or salvage setting as long as >= 6 months from discontinuation have elapsed at the time of randomization
* Progression based on the following criteria:

  * PSA progression: For patients with prior radical prostatectomy (+/- radiation), PSA progression defined by a minimum of two rising PSA levels with an interval of at least 1 week between each determination and a PSA of >= 0.5 ng/ml at screening. For patients with only prior definitive radiation of the prostate, PSA recurrence is defined as PSA >= nadir+2 ng/mL
  * PSA doubling time of =< 12 months at the time of study entry. Calculation of PSA doubling time should include the use of all available PSA values obtained within past 12 months prior to randomization, with a minimum of 3 values >= 0.1 ng/mL PSA values obtained prior to localized therapy will be excluded. PSA doubling time to be estimated using Memorial Sloan Kettering Cancer Center online calculator
  * Identification of up to 5 metastatic lesions or/and pelvic node recurrent sites by advanced imaging technology (PSMA PET/CT or fluciclovine PET/CT). In case of inconsistency between the two imaging modalities, up to 5 lesions in the PSMA/PET will be accepted. All sites should be eligible to be treated with definitive intent. At least one of these lesions will be histologically confirmed. Symptomatic metastatic disease or disease impending symptoms (e.g. brain metastasis, painful bone metastasis, and spine disease) can be treated with definitive local therapy prior to enrollment. This lesion will be counted towards the total number of metastatic lesions
* Must be able to receive luteinizing hormone-releasing hormone (LHRH) agonist or antagonist during the course of the study
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1
* Must be able to swallow tablets
* To avoid risk of drug exposure through the ejaculate (even men with vasectomies), patients must agree while on study drug and for 3 months following the last dose of study drug to:

  * Use a condom during sexual activity
  * Not donate sperm
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 9.0 g/dL
* Platelet count >= 75 x 10^9/L
* Serum albumin >= 3 g/dL
* Calculated creatinine clearance >= 40 mL/min using the Cockcroft-Gault equation
* Serum total bilirubin =<1.5 x upper limit of normal (ULN) or direct bilirubin =< 1.5 x ULN (Note: in subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin, and if direct bilirubin is =< 1.5 x ULN, subject may be eligible)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3.0 x ULN
* Testosterone > 150 ng/dL. For patients treated with ADT with or without short-term first generation anti androgens (e.g. bicalutamide) up to 4 weeks prior to randomization, a testosterone measurement prior to the ADT treatment will be used to determine eligibility, and must have been > 150 ng/dL. If no testosterone level is available from before luteinizing hormone-releasing hormone analogue (LHRHa) injection and within 6 weeks of randomization, the patient will be ineligible

Exclusion Criteria:

* Histologically confirmed recurrence in a prior definitively irradiated prostate cancer field per the judgment of the investigator
* Ongoing androgen deprivation therapy (with or without short-term first generation anti-androgens) for > 4 weeks at the time of randomization
* =< 30 days prior to cycle 1 day 1, patient had:

  * A transfusion (platelets or red blood cells)
  * Hematopoietic growth factors
  * An investigational agent (=< 30 days or 5 half-lives, whichever is longer)
  * Major surgery
* Active hematologic or solid malignancy other than prostate cancer with at least 30% chance of recurrence per investigator assessment; (exceptions: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission)
* Known allergies, hypersensitivity, or intolerance to apalutamide or LHRH agonist/antagonist or excipients
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
* Corrected QT interval by the Fridericia correction formula (QTcF) > 450 msec on the screening electrocardiogram (ECG)
* History of clinically significant cardiovascular disease including, but not limited to:

  * Myocardial infarction or unstable angina =< 3 months prior to treatment initiation
  * Clinically significant cardiac arrhythmia
  * Pulmonary embolism, stroke =< 3 months prior to treatment initiation
  * Congestive heart failure (New York Heart Association class III-IV)
* Known evidence of an active infection requiring systemic therapy such as human immunodeficiency virus (HIV), active hepatitis, or fungal infection
* History of seizure disorder
* Patients receiving medications known to lower the seizure unless discontinued or substituted at least 4 weeks prior to study entry. These medications include:

  * Aminophylline/theophylline,
  * Atypical antipsychotics (e.g., clozapine, olanzapine, risperidone, ziprasidone),
  * Bupropion,
  * Lithium,
  * Meperidine and pethidine,
  * Phenothiazine antipsychotics (e.g., chlorpromazine, mesoridazine, thioridazine),
  * Tricyclic and tetracyclic antidepressants (e.g., amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine)
* Any contraindication that precludes use or radiotherapy for identified lesion treatment per the judgment of the investigator
* Any condition for which, in the opinion of the investigator, participation would not in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Time to prostate specific antigen (PSA) recurrence | From treatment start with androgen deprivation therapy plus apalutamide until PSA recurrence (> 0.2 ng/ml) for patients who received surgery, or PSA >= nadir+2ng/mL for patients who received only prior definitive radiation of the prostate, up to 4 years
  Will estimate with the 95% Bayesian credible interval.

SECONDARY OUTCOMES:
Time to testosterone recovery | From treatment start until testosterone > 150ng/dL, assessed up to 4 years
  Measured using the Kaplan-Meier method.
Eugonadal time to PSA recurrence | Up to 4 years
  Defined as the time to PSA recurrence following testosterone recovery (> 150 ng/dL). Measured using the Kaplan-Meier method.
Overall survival | Up to 4 years
  Measured using the Kaplan-Meier method.
Incidence of adverse events | Up to 4 weeks after last dose of apalutamide
  Safety data will be summarized by treatment arm, category, grade and attribution. Measured by grade 2 or higher adverse events by Common Terminology Criteria for Adverse Events version 5.0.
Time to first new metastasis or local/pelvic recurrence | Up to 4 years
Patient reported outcomes (PRO) | Up to 4 years
  Patient reported outcomes assessed using the following questionnaires EuroQOL 5 Dimensional Questionnaire (EQ-5D-5L) - EuroQOL 5 Dimensional Questionnaire (EQ-5D-5L); Outcome measure is the index value. Range: -0.573 to 1.
Patient reported outcomes (PRO) | Up to 4 years
  Patient reported outcomes assessed using the following questionnaires European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLC-C30): Outcome measure is a raw score, ranging from 0-100.
Patient reported outcomes (PRO) | Up to 4 years
  Patient reported outcomes assessed using the following questionnaires European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire EORTC QLQ-ELD14 Outcome measure is a raw score, ranging from 0-100
Patient reported outcomes (PRO) | Up to 4 years
  Patient reported outcomes assessed using the following questionnaires Expanded Prostate Cancer Index Composite (EPIC-26): Results are presented in a standardized 0-100 scale.
Metabolic syndrome changes | Up to 4 years
  Laboratory parameters that will be measured during screening and active treatment (Lipid panel, blood sugar, HbA1c, Vitamin D, TSH, Testosterone, c-peptide, leptin) as well as measurements of weight and height and bone density measurement results will be used to evaluate changes in parameters predisposing to metabolic syndrome. .Laboratory parameters that will be measured during screening and active treatment (Lipid panel, blood sugar, HbA1c, Vitamin D, TSH, Testosterone, c-peptide, leptin) as well as measurements of weight and height and bone density measurement results
Change in bone density | Up to 4 years
  The results from bone density scanning (DXA scan) will be used to evaluate changes in bone density in the patient population
Imaging changes | Up to 4 years
  Association of changes between baseline and repeat advanced imaging with outcome will be performed, as well as comparison between fluciclovine and PSMA PET/CT modalities, including detection rates and correlation of detected disease volume at baseline with outcome. These changes will be evaluated in correlation with molecular characteristics explored through interrogation of archival and recurrent tissue samples , exosome, steroid and androgen metabolism. Association of changes between baseline and repeat advanced imaging with outcome will be performed, as well as comparison between fluciclovine and PSMA PET/CT modalities, including detection rates and correlation of detected disease volume at baseline with outcome. These changes will be evaluated in correlation with molecular characteristics explored through interrogation of archival and recurrent tissue samples , exosome, steroid and androgen metabolism.
Fluciclovine positron emission tomography/computed tomography (PET/CT) modality assessment | Up to cycle 4, day 1 (each cycle = 28 days)
  Will estimate lesion detection rate based on fluciclovine and prostate-specific membrane antigen (PSMA) PET/CT modalities and the agreement between fluciclovine and PSMA PET/CT results will be assessed through McNemar test.
PSMA PET/CT modality assessment | Up to cycle 4, day 1 (each cycle = 28 days)
  Will estimate lesion detection rate based on fluciclovine and PSMA PET/CT modalities and the agreement between fluciclovine and PSMA PET/CT results will be assessed through McNemar test.

OTHER OUTCOMES:
Identification of response or resistance markers | Up to 4 years
  Identification of markers of response or resistance through correlation with outcomes (interrogation of archival and recurrent tissue samples, exosome, steroid and androgen metabolism)

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Efstathiou, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org